CLINICAL TRIAL: NCT04135742
Title: Effects of Transcranial Alternating Current Stimulation(tACS) Combined With Computerized Cognitive Training for Patients With Mild Cognitive Impairment(MCI)
Brief Title: Effects of tACS Combined With CCT for Patients With MCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Yangpu District Central Hospital Affiliated to Tongji University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-24R
Record Dates: First submitted 2019-10-20; First posted 2019-10-23 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Mild Cognitive Impairment
Keywords: Transcranial Alternating Current Stimulation; Computerized Cognitive Training
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Transcranial Direct Current Stimulation; Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- active tACS+ Cognitive Training group (Experimental): Subjects will receive CCT for a period of 3 months, 24 times, twice a week for 20 minutes each time.
  Placement of stimuli electrodes will be: a) active electrode over the left DLPFC (F3), and b) reference electrode over the right parietal region (P4). The exact location of electrodes will be determined by the 10/20 EEG method with EEG cap. Subjects will have 24 tACS sessions for three months, twice a week.The active tACS group will be stimulated with a 2 mA,40Hz current for 20 minutes each time during the stimulation.
  Interventions: Device: Transcranial Alternating Current Stimulation; Behavioral: Cognitive Training
- sham tACS+Cognitive Training group (Sham Comparator): Subjects will receive CCT for a period of 3 months, 24 times, twice a week for 20 minutes each time.
  Placement of stimuli electrodes will be: a) active electrode over the left DLPFC (F3), and b) reference electrode over the right parietal region (P4). The exact location of electrodes will be determined by the 10/20 EEG method with EEG cap. Subjects will have 24 tACS sessions for three months, twice a week.The sham tACS group will have stimulation lasting only 40 seconds though the electrodes will remain in place for 20 min.
  Interventions: Behavioral: Cognitive Training
- active tACS+ sham Cognitive Training group (Sham Comparator): Subjects will watch neutral pictures on iPad for a period of 3 months, 24 times, twice a week for 20 minutes each time.
  Placement of stimuli electrodes will be: a) active electrode over the left DLPFC (F3), and b) reference electrode over the right parietal region (P4). The exact location of electrodes will be determined by the 10/20 EEG method with EEG cap. Subjects will have 24 tACS sessions for three months, twice a week.The active tACS group will be stimulated with a 2 mA,40Hz current for 20 minutes each time during the stimulation.
  Interventions: Device: Transcranial Alternating Current Stimulation

INTERVENTIONS:
Device: Transcranial Alternating Current Stimulation — Transcranial alternate current stimulation (tACS) is a method of alternative current stimulation that can modulate neural activity by imposing local oscillatory activity.
  Arms: active tACS+ Cognitive Training group; active tACS+ sham Cognitive Training group
Behavioral: Cognitive Training — Cognitive training includes memory, reasoning, processing speed and role playing, etc.
  Arms: active tACS+ Cognitive Training group; sham tACS+Cognitive Training group

SUMMARY:
This goal of this study is to explore the effects of transcranial alternating current stimulation(tACS) combined with computerized cognitive training(CCT) on improving cognition for patients with mild cognitive impairment(MCI). The study will recruit 195 patients with MCI. Participants will undergo baseline cognitve assessment, EEG and structural and functional MRI. Participants will be randomized to active tACS+CCT group, sham tACS+CCT group and active tACS+sham CCT group. At the end of the intervention, 3-month, 6-month and 12-month follow-up, all subjects will repeat the baseline assessments.

DETAILED DESCRIPTION:
tACS is a non-invasive brain stimulation technique that uses a low-intensity alternating current (1 to 2 mA) to apply a sinusoidal current to the scalp, directly interacting with the oscillating cortical activity at a given frequency with a given stimulus intensity. Studies have shown that simultaneous tACS on the left prefrontal lobe and left temporal lobe can significantly improve working memory in healthy older adults. The 40 Hz tACS is gamma oscillation, and more and more studies have pointed out that gamma oscillation regulation disorder is associated with impaired working memory function.CCT can improve the cognition in patients with MCI. We hypothesized that tACS combined with CCT can produce synergistic effects in sensitive brain areas.

ELIGIBILITY:
Inclusion Criteria:

* (1)age ≥ 60 years old with memory impairment; (2) the memory test scores are lower 1.5 SD than the normal control; (3) in addition to memory impairment, other cognitive functions remain relatively intact or only slightly impaired; (4) normal daily living ability; (5) can not reach the diagnostic criteria for dementia, Clinical Dementia Rating (CDR) is 0.5

Exclusion Criteria:

* (1) serious medical diseases such as hypertension, heart disease, severe liver disease, etc.; (2) central nervous system diseases such as cerebrovascular diseases, infectious encephalopathy, brain tumors, etc.; (3) severe depression, schizophrenia and patients who have taken psychotropic substances for a long time; (4) Alzheimer's disease and vascular dementia; (5) history of alcohol dependence and other psychoactive substance abuse; (6) patients with contraindications for magnetic resonance imaging; (7) cannot complete the cognitive function tests for various conditions

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2019-11-11 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline RBANS, Color Word Stroop Test (CWST),Visual Reasoning and Trails Making Task. | up to 3 months(end of the intervention)
  Global cognition will be assessed by the Repeatable Battery for the Assessment of Neuropsychological Status Total Score (RBANS).CWST mainly can examine the executive function. Visual Reasoning will be assessed by the Cambridge Mental Disorders of the Elderly Examination Visual Reasoning Test.Executive function will be assessed by Trails Making Task.
Neuroimage change from baseline Magnetic Resonance Imaging (MRI) | up to 3 months(end of the intervention)
  Including T1, resting state functional MRI, task based functional MRI and Diffusion Tensor Imaging(DTI)
changes in Gamma oscillation intensity (40-80 Hz) over DLPFC | up to 3 months(end of the intervention)
  measured by electroencephalogram (EEG)

SECONDARY OUTCOMES:
Changes from baseline RBANS | 3 months after the end of the intervention,6 months after the end of the intervention and 12 month after the end of the intervention
  Global cognition will be assessed by the Repeatable Battery for the Assessment of Neuropsychological Status Total Score (RBANS).
Changes from baseline Color Word Stroop Test (CWST) | 3 months after the end of the intervention,6 months after the end of the intervention and 12 month after the end of the intervention
  CWST mainly can examine the executive function. There are age-, sex-, and educational year-stratified norms; individuals' z-score can be calculated.
Changes from baseline Visual Reasoning | 3 months after the end of the intervention,6 months after the end of the intervention and 12 month after the end of the intervention
  Visual Reasoning will be assessed by the Cambridge Mental Disorders of the Elderly Examination Visual Reasoning Test.
Changes from baseline Trails Making Task | 3 months after the end of the intervention,6 months after the end of the intervention and 12 month after the end of the intervention
  Executive function will be assessed by Trails Making Task.
Changes from baseline Geriatric Depression Scale (GDS) | up to 3 months(end of the intervention),3 months after the end of the intervention,6 months after the end of the intervention and 12 month after the end of the intervention
  The Geriatric Depression Scale will be used to measure neuropsychiatric symptoms. It ranges from 0 to 30, and higher value represents a worse outcome.
Changes from baseline in Geriatric Anxiety Inventory (GAI) | up to 3 months(end of the intervention),3 months after the end of the intervention,6 months after the end of the intervention and 12 month after the end of the intervention
  Geriatric Anxiety Inventory (GAI) will be used to measure neuropsychiatric symptoms.
Neuroimage changes from baseline Magnetic Resonance Imaging (MRI) | 6 months after the end of the intervention and 12 month after the end of the intervention
  Including T1, resting state functional MRI, task based functional MRI and Diffusion Tensor Imaging(DTI)
Side-effects of tACS | At each stimulation session,up to 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Chunbo Li, Ph.D, Principal Investigator — Shanghai Mental Health Center
Locations (2):
- China (2):
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality
  - Yangpu District Central Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No